Title: Comparison of obturator nerve blockade and neuromuscular blockade for the prevention of adductor spasm in patients undergoing transurethral resection of bladder tumors.

NCT: NCT03063255

Date: October 25, 2018



#### VA RESEARCH CONSENT FORM



| Subject Name: | | Date | |
|---|---|---|---|
| | n of obturator nerve blockade ar<br>tor spasm in patients undergoin | | |
| Principal Investigator: José R | Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |
| UF Institut | ional Review Board<br>SITY of FLORIDA | | |
| | CONSENT FORM<br>ate in Research | | |
| | Introdu | CTION | |
| Name of person see | king your consent:t & position: | | |

Please read this form which describes the study in some detail. A member of the research team will also describe this study to you and answer all of your questions. Your participation is entirely voluntary. If you choose to participate you can change your mind at any time and withdraw from the study. You will not be penalized in any way or lose any VA or other benefits to which you would otherwise be entitled if you choose not to participate in this study or to withdraw. If you have questions about your rights as a research subject, concerns, complaints, wish to discuss problems or talk to someone independent of the research staff, obtain information, or offer input, please call either of the following offices: (1) the University of Florida Institutional Review Board (IRB) office at (352) 273-9600; or (2) the North Florida/South Georgia Veteran's Health System Research Service Office at (352) 548-6069.

IRB Project #: 201601962 IRB Version: 04/25/2015 PI Version: 10/13/2018

| 人 | Y | T | Department of Veterans Affairs |
|---|----|----------|--------------------------------|
| 7 | 77 | <b>y</b> | Department of Veterans Affairs |

#### VA RESEARCH CONSENT FORM

| ARB-01 | Appro |
|---------------|----------|
| D ed | ed U |
| Joseph Joseph | 10 841.2 |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and neuromus adductor spasm in patients undergoing transureth | | |
| | ator: _José R. Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |

## **GENERAL INFORMATION ABOUT THIS STUDY**

1. Name of Participant ("Study Subject")

For PI Use:

Participant Social Security Number:

SSN should be written on this consent form by the research team prior to scanning into the VHA health record; if the subject does not have a VHA health record, this requirement is N/A.

## 2. What is the Title of this research study?

Comparison of obturator nerve blockade and neuromuscular blockade for the prevention of adductor spasm in patients undergoing transurethral resection of bladder tumors

3. Who can you call if you have questions, concerns, or complaints about this research study?

Principal Investigator: José R. Soberón, Jr, MD

Department of Anesthesiology NF/SG Veterans Health System 1601 Archer Road

Gainesville, Florida 32608 Pager: (352) 413-2317

## 4. Who is paying for this research study?

The sponsor of this study is Veterans Administration

## 5. Why is this research study being done?

Agreeing to become involved in any research is always voluntary. By signing this form, you are not waiving any of your legal rights. If you decide not to participate in this

IRB Project #: 201601962 IRB Version: 04/25/2015 PI Version: 10/13/2018

 **VA Form 10-1086** 



#### VA RESEARCH CONSENT FORM



| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and<br>adductor spasm in patients undergoing | | • |
| | r: José R. Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |

research, you will not be penalized in any way and you will not lose any benefits to which you are entitled. If you have questions about your rights as a research subject, please call the University of Florida Institutional Review Board (IRB) office at (352) 273-9600 or the North Florida/South Georgia Veteran's Health System Research Service Office at (352) 548-6069.

- a) In general, what is the purpose of the research, how long will you be involved? The purpose of this research study is to compare two techniques to prevent the obturator reflex in patient undergoing transurethral resection of a bladder tumor (TURBT). You will be involved until you receive the follow-up phone call 24-48 hours after surgery.
- b) What is involved with your participation, and what are the procedures to be followed in the research?

The obturator nerve runs next to the bladder and surgery on the bladder sometimes makes the nerve move the leg while you are under anesthesia. This is called the obturator reflex. An obturator nerve block is performed to block the nerve from making the leg move. General anesthesia with muscle relaxants have also been used to prevent leg movement but the two techniques have never been directly compared.

A nerve block involves injecting numbing medications around a nerve to decrease leg movement during surgery. An ultrasound machine is used to help see the nerve before injecting the numbing medicine. When an ultrasound machine is used during a block it is called an ultrasound-guided block.

You are being asked to be in this research study because you are scheduled to have a TURBT.

- c) What are the likely risks or discomforts to you?
  - Because the nerve block is performed after you are under general anesthesia, there is no additional discomfort from the study interventions.
- d) What are the likely benefits to you or to others from the research?
   Potential benefits include prevention of the obturator reflex. The information

obtained from this study may help providers decide on the best approach to prevent the obturator reflex in future surgeries.

IRB Project #: 201601962 IRB Version: 04/25/2015 PI Version: 10/13/2018  VA Form 10-1086

| Department of Veterans Affa | fai |
|-----------------------------|-----|
|-----------------------------|-----|

#### VA RESEARCH CONSENT FORM

| (IRB | ,01 A <sub>A</sub> | Prop |
|------|--------------------|------|
| | П | ed 2 |
| oto. | QA 10 | ET. |
| 4 | OI AD | 4. |

| Subject Name: _ | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and neurom adductor spasm in patients undergoing transure | | |
| Principal Investig | ator: José R. Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |

e) What are the appropriate alternative procedures or courses of treatment, if any, that might be helpful to you?

You will likely receive general anesthesia, muscle relaxant medications, and/or an obturator nerve block for your surgery regardless of your decision to participate in the research study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Additional and more detailed information is provided within the remainder of this Informed Consent form, please read before deciding if you wish to participate in this study.

#### WHAT CAN YOU EXPECT IF YOU PARTICIPATE IN THIS STUDY?

6. What will be done as part of your normal clinical care (even if you did not participate in this research study)?

Normal clinical care is medical or other treatment or services that you would receive even if you did not participate in this research study. You will receive general anesthesia for your procedure as well as a obturator nerve or muscle relaxing medications regardless of whether or not you choose to participate in the study.

7. What will be done only because you are in this research study?

If you agree to be in this study, we will ask you to do the following things:

You will be asked to stand from a chair, walk 10 feet, and return to the seated position. A device measuring muscle strength will be used to record the strength in your legs. The device measures your strength by having you push against it with your leg. It is not associated with discomfort.

Your surgery will be performed as per normal standard of care. If you agree to participate in this study you will be randomized to 1 of 2 groups. Once consent is obtained, enrollees will be randomly allocated by computer-generated randomization to one of the study groups. Randomization is like a flip of a coin that


| Department of Veterans Affa |
|-----------------------------|
| Department of Veterans And |

#### VA RESEARCH CONSENT FORM

| A P | 3.01 A | PPO |
|-------|---------|------|
| D po | | ed U |
| -0,70 | 10 A 10 | BAI. |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and adductor spasm in patients undergoing to | | |
| | | | North Florida/South Georgia |
| Principal Investiga | ator: José R. Soberón, Jr., MD | VAMC: | Veterans Health System |

will determine to which group you will be assigned. Both techniques are currently in use at this facility.

The nerve block or muscle relaxing medications will be administered while you are under anesthesia. You will then have your surgery. You will receive the nerve block or muscle relaxing medications even if you do not agree to be in this study. Three stickers will be placed on your thigh and they will be connected to a machine that measures muscle activity to determine leg movement during your procedure.

Medications given during surgery and in the recovery room will be recorded. One hour after arrival to the recovery room or when you are ready for discharge, we will ask you to repeat the same evaluation as before (walking and measuring your leg strength).

You will be called 24-48 hours after surgery to see if there were any complications with your procedure.

The Principal Investigator listed in question 3 of this form and the research team conducting the research procedures described above will monitor how you do during the research. If you have any questions about the research procedures now or at any time during the study, please contact one of the research team members listed in question 3 of this form.

Once this research study is completed, any information that could identify you might be removed from any identifiable private information or identifiable biospecimens collected and that, after such removal, the information or biospecimens could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

If you have any questions now or at any time during this Research Study, please contact one of the Research Team members listed in question 3 of this form.

## 8. How long will you be in this research study?

Your participation will be complete after the follow-up phone call(s) or 3 days, whichever happens first.

#### 9. How many people are expected to take part in this research study?

70.


| 5 | $\mathbf{Z}$ | Department of Veterans Affai |
|---|--------------|------------------------------|
|---|--------------|------------------------------|

#### VA RESEARCH CONSENT FORM

| 3 | B-01 | $A_{P_{i}P_{i}}$ | ro, |
|------|------|------------------|------|
| d U | IJ | F | ed L |
| al O | ddy | . 0 | E E |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade ar<br>adductor spasm in patients undergoin | | |
| Principal Investiga | ator: José R. Soberón Jr. MD | North Florida/ | 0 |

# WHAT ARE THE RISKS AND BENEFITS OF THIS STUDY AND WHAT ARE YOUR OPTIONS?

## 10. What are the possible discomforts and risks from taking part in this research study?

Both the nerve block and muscle relaxing medications are commonly performed and acceptable techniques to prevent obturator spasm. These (nerve block or muscle relaxants) will be administered while you are under general anesthesia, so no additional discomfort should be expected. Risks of the nerve block may include nerve damage, intravascular injection of local anesthetic, cardiac arrest, seizure, bleeding/hematoma, infection, ineffective or failed block, pain at the injection site, or numbness or tingling (paresthesia). To date, no complications have been reported or associated with the obturator nerve block.

Risks of muscle relaxing medications may include weakness, fatigue, and difficulty breathing, which may require keeping the breathing tube in place after surgery. Other risks may include pulmonary aspiration (acid from the stomach comes up into the lungs) and longer time spent in the recovery room.

Adhesive electrodes (stickers) will be placed on your leg during surgery to measure leg muscle movement while you are asleep. Very rarely, skin irritation may occur at the site of placement. This generally goes away in 2-3 days (or less).

Researchers will take appropriate steps to protect any information they collect about you. However there is a slight risk that information about you could be revealed inappropriately or accidentally. Depending on the nature of the information such a release could upset or embarrass you, or possibly even affect your insurability or employability.

Other possible risks to you may include: Because we are asking you to stand up and walk before and after your procedure, there is a possibility of falling. Every possible precaution, including a fall prevention belt and close supervision, will be taken to minimize risk of falling. The device that measures your strength by having you push against it with your leg is not associated with discomfort.

This study may include risks that are unknown at this time.

Participation in more than one research study or project may further increase the risks to you. If you are already enrolled in another research study, please inform one of the


| Department of Veterans Aff | 1 | W | Department of Veterans Affa |
|----------------------------|---|---|-----------------------------|
|----------------------------|---|---|-----------------------------|

#### VA RESEARCH CONSENT FORM

| RB-01 | Appro |
|--------|----------|
| r<br>P | ed U |
| orday | 10 BAL 2 |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and neuro<br>adductor spasm in patients undergoing transul | | • |
| Principal Investigato | r: José R. Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |

research team members listed in question 3 of this consent form or the person reviewing this consent with you before enrolling in this or any other research study or project.

Throughout the study, the researchers will notify you of any new information that may become available and might affect your decision to remain in this study. This includes, but is not limited to, information that may affect your safety, well-being or medical care.

If you wish to discuss the risks or discomforts described above or any discomforts you may experience, please ask questions now or call one of the research team members listed in question 3 of this form.

#### 11a. What are the potential benefits to you for taking part in this research study?

Because the obturator reflex may interfere with tumor resection, performance of an obturator block or use of neuromuscular relaxing agents may block the reflex and allow for safer operating conditions and improved cancer removal.

Leg strength and fall risk assessments will be performed for all patients to determine suitability for discharge. At the present time, there are no data regarding fall risk in patients with obturator blocks. Evaluating leg strength and ability to walk may help determine if it is safe for you to be discharged from the hospital if you receive an obturator block.

## 11b. How could others possibly benefit from this study?

This study will help future anesthesia providers decide which technique (nerve block or muscle relaxants) is better for preventing obturator spasm. The success rate and safety of one approach versus the other is not known. The results of this study may be used to guide clinical decisions for future patients undergoing TURBT or to conduct larger prospective studies.

## 11c. How could the researchers benefit from this study?

In general, presenting research results helps the career of a scientist. Therefore, the Principal Investigator listed in question 3 may benefit if the results of this study are presented at scientific meetings or in scientific journals.


| Department of Veterans Affair |
|-------------------------------|
| Department of Veterans Affair |

#### VA RESEARCH CONSENT FORM

| TRB. | $MA_{P_{D_{r_{O_{A}}}}}$ |
|------|--------------------------|
| Î | TF ed ~ |
| orda | TEN OF THE |
| - 'Q | A 1010 |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade ar<br>adductor spasm in patients undergoin | | • |
| Title of olday. | | North Florida/South Georgia<br>Veterans Health System | |

#### 12. What other choices do you have if you do not want to be in this study?

A nerve block or muscle relaxants will be administered in an attempt to minimize obturator spasm whether you choose to participate in the study or not.

#### 13a. Can you withdraw from this study?

You are free to withdraw your consent and to stop participating in this study at any time. If you do withdraw your consent, you will not be penalized in any way and you will not lose any benefits to which you are entitled.

If you decide to withdraw your consent to participate in this study for any reason, please contact one of the research team members listed in question 3 of this form. They will tell you how to stop your participation safely.

If you have any questions regarding your rights as a research subject, please call the Institutional Review Board (IRB) office at (352) 273-9600.

## 13b. If you withdraw, can information about you still be used and/or collected?

If you withdraw from this study, your research information will no longer be collected. However, information that has already been collected will continue to be used to the extent that the researchers have used it in this research study.

## 13c. Can the Principal Investigator withdraw you from this study?

You may be withdrawn from the study without your consent for the following reasons:

- the study doctor thinks it necessary for your health or safety;
- you have not followed study instructions;
- the sponsor has stopped the study; or
- administrative reasons require your withdrawal.


| Department of Veterans Affai |
|------------------------------------|
| <br>Dopartinonic or votorano / ina |

#### VA RESEARCH CONSENT FORM

| 4 | RB-01. | $Ap_{D_{r_{O}}}$ | |
|-----|---------|------------------|-------|
| 0 1 | TT | | pod / |
| 9 | Proddy. | | 4 |
| | AGA | 10 80 | |

| Subject Name: | | Date |
|---|---|---|
| Title of Study: | • | nd neuromuscular blockade for the prevention of<br>g transurethral resection of bladder tumors |
| Principal Investig | uator: José R. Soberón, Jr., MD | North Florida/South Georgia |

#### WHAT ARE THE FINANCIAL ISSUES IF YOU PARTICIPATE?

#### 14. If you choose to take part in this research study, will it cost you anything?

There will be no costs to you for any procedure, treatment or testing done as part of this research study. However, medical care and services provided by the VA that are not being done only for this study (e.g., normal hospital and prescription expenses which are not part of the research study) will be charged to you or your insurance. These costs may not be charged if you are a veteran and you are being treated at the North Florida/South Georgia Veterans Health System (NF/SG VHS), however some Veterans are required to pay co-payments for medical care and services provided by the VA. These co-payment requirements will continue to apply to VA-provided medical care and services that are not part of this study."

#### 15. Will you be paid for taking part in this study?

No.

## 16. What if you are injured because of the study?

If you experience an injury or illness as a result of your participation in this VA approved research study, all medical treatment considered necessary by your physician (emergency as well as medical treatment beyond emergency) will be provided by the VA. There will be no cost to you, unless you fail to follow the directions of the study procedures. Care will be provided at a VA medical facility unless the VA medical facility is not capable of providing the care. If this occurs, you will be treated by a private facility or physician and the VA will pay the private facility or physician for the reasonable cost of your care. In some cases the VA may approve private care for a non-veteran.

If you do not follow study procedures, you may be treated by the VA on the basis of your veteran's eligibility. If you are not a veteran and have not followed study procedures the VA can only provide limited care at your expense.

No additional money has been set aside for pain, suffering or any money losses you may suffer during your treatment. You have not waived any legal rights by signing this form.


| (X) | Department of Veterans Affa |
|-----|-----------------------------|
| | Department of Veterans And |

#### VA RESEARCH CONSENT FORM

| A IRB- | $^{11}A_{P_{p_{r_{o_{h}}}}}$ |
|---|---|
| P. | |
| ordd | THE STATE OF THE S |
| qQ | A 10 0 |

| Subject Name: | | Date | |
|---|---|---|---|
| Title of Study: | Comparison of obturator nerve blockade and neuromuscular blockade for the prevention of adductor spasm in patients undergoing transurethral resection of bladder tumors | | |
| Principal Investigato | r: José R. Soberón, Jr., MD | VAMC: | North Florida/South Georgia<br>Veterans Health System |

In the event of a research-related injury, have questions about any discomforts that you experience while participating in this study or if you experience an adverse reaction, please immediately contact the Principal Investigator listed in question 3 of this form during the day and 786-247-2749 after business hours. If you seek emergency hospitalization in a private hospital because you are unable to come to the VA, have a family or friend contact your study doctor so that the VA can coordinate care with the private hospital.

## 17. How will your privacy and the confidentiality of your research records be protected?

Information collected about you will be stored in locked filing cabinets or in computers with security passwords. Only certain people have the legal right to review these research records, and they will protect the secrecy (confidentiality) of these records as much as the law allows. These people include the researchers for this study, certain University of Florida officials, the hospital or clinic (if any) involved in this research, and the Institutional Review Board (IRB; an IRB is a group of people who are responsible for looking after the rights and welfare of people taking part in research). Certain federal agencies such as the Office for Human Research Protections (OHRP), the VA Office of Research Oversight (ORO), or the VA Office of the Inspector General (OIG), that oversee human subject research may also have the legal right to review your records. Otherwise your research records will not be released without your permission unless required by law or a court order.

Researchers will take appropriate steps to protect any information they collect about you. However there is a slight risk that information about you could be revealed inappropriately or accidentally. Depending on the nature of the information such a release could upset or embarrass you, or possibly even affect your insurability or employability.

If the results of this research are published or presented at scientific meetings, your identity will not be disclosed.


| <b>(2)</b> | Department of Veterans Affairs |
|------------|--------------------------------|

## **VA RESEARCH CONSENT FORM**

Date

| Subject Name | Posts. |
|---|---|
| • | Date ade and neuromuscular blockade for the prevention of ergoing transurethral resection of bladder tumors |
| Principal Investigator: José R. Soberón, Jr., MD | North Florida/South Georgia VAMC: Veterans Health System |
| SIGNATURES | |
| As an investigator or the investigator's representative, I have explained to the participant the purpose, the procedures, the possible benefits, and the risks of this research study; the alternatives to being in the study; and how privacy will be protected: | |
| Signature of Person Obtaining Consent | Date |
| You have been informed about this study's purpose, procedures, possible benefits, and risks; the alternatives to being in the study; and how your privacy will be protected. You have received a copy of this Form. You have been given the opportunity to ask questions before you sign, and you have been told that you can ask other questions at any time. | |
| You voluntarily agree to participate in this any of your legal rights. | study. By signing this form, you are not waiving |

IRB Project #: 201601962 IRB Version: 04/25/2015 PI Version: 10/13/2018

Signature of Person Consenting